CLINICAL TRIAL: NCT00769457
Title: OptiLink HF Study (Optimization of Heart Failure Management Using Medtronic OptiVol® Fluid Status Monitoring and Medtronic CareLink® Network)
Brief Title: OptiLink HF Study: Optimization of Heart Failure Management Using Medtronic OptiVol Fluid Status Monitoring and CareLink Network
Acronym: OptiLink-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEN_G_CA_8
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2016-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Arm with activated OptiVol / Carelink-system, event-triggered physician alert and physician access to Cardiac Compass data
  Interventions: Device: Access Arm
- 2 (No Intervention): Arm with standard ICD - CRT-D therapy, no OptiVol and no Carelink

INTERVENTIONS:
Device: Access Arm — Active OptiVol-System with CareAlert via CareLink
  Other Names: Medtronic CRT-D and ICD-VR / DR with OptiVol, Conexus-Telemetry, CareLink:; Concerto , Consulta , Virtuoso , Secura , Protecta XT
  Arms: 1

SUMMARY:
Patients suffering from heart failure and a markedly reduced pumping capacity and sometimes desynchronization of the lower chambers of the heart have a higher risk of suffering sudden cardiac death.

These patients can be treated with an Implantable Cardiac Defibrillator that terminates dangerously fast heartbeats and in case of asynchronous pumping of the heart can also re-synchronize the lower chambers of the heart (ICD- or CRT-D-system). Patients that moreover suffered from a worsening of their cardiac status (cardiac decompensation) and had to be hospitalized for this reason have a higher risc to have following decompensations. New technology, incorporated into modern Medtronic ICD- and CRT-D-Systems, that measures the amount of water in the lungs is able to warn before such a dangerous worsening occurs. If coupled with modern data transmitting technology (CareLink), automatic information in case of a worsening of the cardiac status can be sent to caregivers, who in turn can react timely in order to prevent a worsening an subsequent hospitalization.

The study examines to which extent this new technology prevents potentially adverse cardiac situations and / or hospitalizations and has an influence of the duration of patient´s lives.

DETAILED DESCRIPTION:
The objective of the study is to establish whether the use of event-triggered HF-disease management through Medtronic's OptiVol® fluid status monitoring with an automatically generated wireless CareAlert® notification of the clinician via the Medtronic CareLink® Network can reduce cardiovascular related hospitalizations and the number of deaths in a subject population with HF and ICD / CRT-D treatment as compared to standard clinical assessment. As a measure for the reduction of hospitalizations and deaths the rate of all cause deaths or cardiovascular related hospitalizations will be determined.

ELIGIBILITY:
Inclusion Criteria

* Subjects have a Medtronic Virtuoso™ ICD single- or dual-chamber or Concerto™ CRT-D or subsequently market released Medtronic device providing at least the same functionality) implanted, including device replacement. Subjects with CRT-D must fulfill CRT-indication as described in the ESC guidelines for cardiac pacing and cardiac resynchronization therapy 2007: EF ≤ 35% and NYHA III, and LVEDD ≥ 55 mm, and QRS ≥ 120 ms, and optimized therapy
* Subjects with stable chronic heart failure (CHF) in New York Heart Association (NYHA) class II or III for at least 30 days and left ventricular ejection fraction of no more than 35% (most recent measurement within 6 months prior to randomization by echocardiography or contrast ventriculography, magnetic resonance or nuclear imaging, based on local practice), on optimal target or maximal tolerated dose of ACE-inhibitors or angiotensin receptor blockers, ß-blockers and diuretics if clinically indicated to reduce fluid retention and one of the following criteria:
* At least one hospitalization due to the heart failure within the last 12 months before enrollment
* Or one course of ambulatory IV-or oral diuretic treatment or a BNP value of > 400 pg/ml or a NT-proBNP values > 450 in subject < 50 years, > 900 (50-75 years) and > 1800 subject of than 75 years old within 30 days of enrollment
* Written informed consent by the subject for study participation prior to clinical investigation plan specific procedures,
* The subject must be able and willing to comply with the clinical investigation plan and willing to remain available for follow-up visits to the study closure,
* Subjects or the subject's caregiver must be willing and able to use the Medtronic CareLink® monitor as instructed and to perform the required duties, if subject is randomized to the access arm.

Exclusion Criteria:

* Subjects with chronic renal failure needing renal dialysis
* Subjects with serum creatinine > 2.5 mg/dl, measured within 14 days prior to enrollment,
* Subjects with severe to very severe Chronic Obstructive Pulmonary Disease (COPD) as determined by physician and documented in medical records (Stage III and Stage IV),
* Subjects with suspected or confirmed COPD require a current test of lung function (not more than 12 months before inclusion). If the "forced expiratory volume" is <1.0 L/sec,the subject may not participate in the study,
* Subjects on the heart transplantation list or subjects with transplanted hearts,
* Subjects listed for valve replacement or interventional valve therapy,
* Subjects with myocardial infarction within the last 40 days before implant. MI is defined by typical changes in biochemical markers including troponin levels > 3 times the upper limits of normal and creatinine kinase < 2 times of upper limit, or with CKMB greater than the upper limit of normal, combined (for all enzymes) with at least one of the following ischemic symptoms, ECG changes consistent of diagnostic ST-T wave changes or pathologic Q waves or new LBBB,
* Subjects with stroke within 40 days prior randomization,
* Subjects who have had a percutaneous coronary intervention within 3 months prior to randomization,
* Subjects with cardiac surgery within 90 days of randomization,
* Subjects with complex and uncorrected Congenital Heart Disease,
* Subject's life expectancy is less than 18 months in the opinion of the physician,
* Subjects in situations that would limit participation, not eligible to receive a CareLink® monitor (e.g. hearing or speech impaired with no family member or caregiver available to assist, or those who spend extended periods abroad, or those who intend to enroll in a study that would preclude use of the monitor),
* Subject is participating in a concurrent intervention study,
* Subject or the subject's caregiver is unwilling to give consent for the release of information for the evaluation or to give additional consent for the release of subject medical and privacy data for CareLink® subjects,
* Subjects with exclusion criteria required by local law (age < 18, women who are pregnant or breastfeeding)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2008-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
All-cause of death or unplanned admission to hospital for cardiovascular reason from day of patient informed consent sign off | 18 Months

SECONDARY OUTCOMES:
Number of HF-related hospitalization during follow-up, HF-related hospitalization, Sum of follow-up days minus days alive and out of the hospital, All cause mortality, Cardiovascular Mortality, | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boehm, Professor, Principal Investigator — Universitätsklinikum des Saarlandes, Homburg-Saar; Johannes Brachmann, Professor, Study Chair — Klinikum Coburg GmbH
Locations (1):
- Universitätsklinikum des Saarlandes, Homburg-Saar, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brachmann J, Bohm M, Rybak K, Klein G, Butter C, Klemm H, Schomburg R, Siebermair J, Israel C, Sinha AM, Drexler H; OptiLink HF Study Executive Board and Investigators. Fluid status monitoring with a wireless network to reduce cardiovascular-related hospitalizations and mortality in heart failure: rationale and design of the OptiLink HF Study (Optimization of Heart Failure Management using OptiVol Fluid Status Monitoring and CareLink). Eur J Heart Fail. 2011 Jul;13(7):796-804. doi: 10.1093/eurjhf/hfr045. Epub 2011 May 8. PMID 21555324
- [Result] Bohm M, Drexler H, Oswald H, Rybak K, Bosch R, Butter C, Klein G, Gerritse B, Monteiro J, Israel C, Bimmel D, Kaab S, Huegl B, Brachmann J; OptiLink HF Study Investigators. Fluid status telemedicine alerts for heart failure: a randomized controlled trial. Eur Heart J. 2016 Nov 1;37(41):3154-3163. doi: 10.1093/eurheartj/ehw099. Epub 2016 Mar 16. PMID 26984864
- See also: Klinik für Innere Medizin III - Kardiologie, Angiologie und internistische Intensivmedizin — http://www.uniklinikum-saarland.de/de/einrichtungen/kliniken_institute/kardiologie